CLINICAL TRIAL: NCT04582435
Title: A Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of Insulin Icodec in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4569; U1111-1244-4346 (Other: World Health Organization (WHO)); 2019-004606-10 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-10-08; First posted 2020-10-09 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insulin icodec (Experimental): Participants will receive individualised weekly doses of insulin icodec
  Interventions: Drug: Insulin Icodec

INTERVENTIONS:
Drug: Insulin Icodec — Participants will receive 1 dose from a prefilled pen, administered subcutaneously (under the skin), once a week by designated study staff, for a total of at least 8 and a maximum of 16 doses which equals 8-16 weeks of treatment.

SUMMARY:
The aim of the study is to improve clinical outcomes for patients with type 2 diabetes by limiting the burden associated with insulin treatment.

Participants will get insulin degludec as well as insulin icodec - Insulin icodec is a new medicine while insulin degludec is commonly used and prescribed by doctors.

Participants will administer subcutaneous injections of insulin degludec once daily for at least one week (7 injections) but this period may be extended up to 8 weeks. Thereafter, once weekly subcutaneous injections of insulin icodec will follow, resulting in a total of at least 8 but not more than 16 subcutaneous injections of icodec.

The study will last for about 17-32 weeks Participants will have at least 5 in-house visits (where participants will stay at the clinic) and 17 outpatient visits with the study doctor.

Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-75 years (both inclusive) at the time of signing informed consent
* Body mass index between 18.0 and 38.0 kg/m^2 (both inclusive)
* HbA1c (glycated haemoglobin) below or equal to 9 percentage (75 mmol/mol) at screening
* Current daily basal insulin treatment greater than or equal to 0.2 (I)U/kg/day with or without any of the following anti-diabetic drugs/regimens with stable doses greater than or equal to 90 days prior to the day of screening: 1) Any metformin formulation 2) Other oral antidiabetic drugs: DPP-4 nhibitors / SGLT2 inhibitors / Oral combination products (for the allowed individual oral antidiabetic drugs)
* Oral or injectable GLP-1 Receptor Agonists

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
AUCIco,τ,SS, Area under the serum insulin icodec concentration-time curve during one dosing interval at steady state | From 0 to 168 hours after trial product administration (Day 50)
  pmol*h/L

SECONDARY OUTCOMES:
AUCGIR,0-36h,SS,Area under the glucose infusion rate-time curve at steady state | From 0 to 36 hours after trial product administration (Day 36)
  mg/kg
AUCGIR,40-64h,SS,Area under the glucose infusion rate-time curve at steady state | From 40 to 64 hours after trial product administration (Day 43)
  mg/kg
AUCGIR,144-168h,SS,Area under the glucose infusion rate-time curve at steady state | From 144 to 168 hours after trial product administration (Day 50)
  mg/kg
AUCGIR,τ,SS,model, Model-based area under the glucose infusion rate-time curve during one dosing interval at steady state | From 0 to 168 hours after trial product administration (Day 50)
  mg/kg
AUCIco,τ,SS, Area under the serum insulin icodec concentration-time curve during one dosing interval at steady state | From 0 to 168 hours after trial product administration (Day 36 and 43)
  pmol*h/L
Dose-normalised AUCIco,τ,SS, Area under the serum insulin icodec concentration-time curve during one dosing interval at steady state divided by dose | From 0 to 168 hours after trial product administration (Day 50)
  (pmol*h/L)/(U/kg)
Cmax,Ico,SS, Maximum observed serum insulin icodec concentration during one dosing interval at steady state | From 0 to 168 hours after trial product administration (Day 36, 43 and 50)
  pmol/L
Dose-normalised Cmax,Ico,SS, Maximum observed serum insulin icodec concentration after the last dose divided by dose | From 0 to 168 hours after trial product administration (Day 50)
  (pmol/L)/(U/kg)
tmax,Ico,SS, Time to maximum observed serum insulin icodec concentration after the last dose | From 0 to 168 hours after trial product administration (Day 50)
  hours
t½,Ico,SS, Terminal half-life for insulin icodec at steady state | Terminal part of the serum insulin icodec concentration-time curve where the curve is well approximated by a straight line on logarithmic scale after last trial product administration (Day 50)
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Pieber TR, Asong M, Fluhr G, Holler V, Kristensen NR, Larsen JH, Ribel-Madsen R, Svehlikova E, Vinther S, Voortman M, Haahr H. Pharmacokinetic and pharmacodynamic properties of once-weekly insulin icodec in individuals with type 2 diabetes. Diabetes Obes Metab. 2023 Dec;25(12):3716-3723. doi: 10.1111/dom.15266. Epub 2023 Sep 11. PMID 37694740